CLINICAL TRIAL: NCT06487780
Title: Evaluating the Feasibility and Acceptability of a Lifestyle Intervention to Prevent Recurrence of Diabetic Foot Ulcers: A Pilot Study
Brief Title: Evaluating a Lifestyle Intervention to Prevent Recurrence of Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Tze-Woei Tan, Associate Professor of Clinical Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APP-24-03267
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer; Foot Ulcer, Diabetic; Foot Wound
Keywords: Diabetic foot ulcer, lifestyle intervention
MeSH Terms: conditions — Diabetic Foot; Foot Injuries | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups, with an equal number in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle-focused Occupational Therapy (OT) Intervention (Experimental): Participants in the intervention group will engage in telemedicine sessions led by trained occupational therapists.
  Interventions: Behavioral: Lifestyle-focused Occupational Therapy Intervention
- Education (Active Comparator): Participants in the control group will receive standard education on foot self-care and offloading treatment aimed at preventing foot ulcer recurrence.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Lifestyle-focused Occupational Therapy Intervention — The proposed intervention, led by trained occupational therapists, will focus on establishing sustainable self-care routines. It will consist of approximately 12 biweekly sessions, each lasting about an hour on average. Therapists will customize session timing and duration based on participant needs.
  Arms: Lifestyle-focused Occupational Therapy (OT) Intervention
Other: Education — Participants in the education group will receive standardized education materials on diabetic foot ulcers (DFUs), foot care, and offloading treatment to prevent foot ulcer recurrence.
  Arms: Education

SUMMARY:
People with diabetes often experience foot ulcers, which can harm their ability to move, lower their quality of life, and increase the chances of losing a limb. These diabetic foot ulcers (DFUs) commonly come back (recur) even after they've healed, so it's crucial to stop them from returning to avoid toe, foot , or leg amputation. While wearing special shoes to reduce pressure on the feet is essential for healing and preventing DFUs, many people struggle to follow this treatment plan once their ulcers have healed. This study aims to see if a lifestyle-focused program can help participants create daily routines and habits that make it easier to consistently use special shoes and take care of their diabetes and feet to prevent ulcers from recurring.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFUs) are a significant complication of diabetes, responsible for 80% of lower extremity amputations in the United States and posing a substantial burden on patients and society. Despite treatment, up to 23% of DFUs remain unhealed at 12 months, with recurrence rates of 40% within a year and 65% within three years. Proper offloading of foot pressure and glucose control is crucial for preventing recurrent DFUs, especially in cases of neuropathy. While standard clinical practice includes patient education and therapeutic footwear prescription, adherence to offloading treatment often falls short due to non-medical factors such as insufficient understanding and difficulties integrating offloading into daily routines. To tackle these challenges, we propose a lifestyle-focused intervention, conducted by trained occupational therapist (OT), aiming at fostering consistent self-care habits and routines.The objective of this pilot trial is to evaluate the feasibility acceptability of a lifestyle-focused OT intervention for enhancing offloading treatment in high-risk individuals with a history of healed DFUs.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 21 years
* Healed diabetic foot ulcer within the past twelve months
* Able to walk independently (use of a cane is acceptable)

Exclusion Criteria:

* Current active diabetic foot ulcer
* History of amputation beside toe or part of the foot
* Non-ambulatory at baseline
* Self-reported deafness/blindness.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants who have completed the study | 6-month
  Investigators will measure participant attendance, completion of planned/scheduled sessions, retention of participants in the intervention and education (control) groups.

SECONDARY OUTCOMES:
Numbers of participants with diabetic foot ulcer recurrence | 6-month
  Rates of foot ulcer recurrence and any amputation.
Numbers of participants who report satisfaction with the program | 6-month
  Participants will complete the Short-form Patient Satisfaction Questionnaire (PSQ-18). The 18 items' scale ranges from 1 (strong agree) to 5 (strongly disagree). Selected participants will be invited to participate in semi-structured interviews.
Number of participants with diabetes distress | 6-month
  Participants will complete the Diabetes Distress Scale (DDS), a 17-item self-report instrument. Each item is rated on a 6-point scale from 1 (not a problem) to 6 (a very significant problem.
Participant's Quality of Life | 6-month
  Participants will complete the Patient-Reported Outcomes Measurement Information System (PROMIS) that evaluate physical, mental, and social health.

CONTACTS AND LOCATIONS:
Overall Officials: Tze Woei Tan, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to share de-identified demographic, clinical, and survey data, along with qualitative data from interviews. This data will be stored in USC-provided OneDrive accounts, approved for Confidential Data storage according to USC standards. All de-identified scientific data, including raw/measured and derived data, will be preserved and shared to support reproducibility and reusability. Research results will be published in peer-reviewed scientific journals and presented at selected scientific meetings. Manuscripts accepted by journals without free access will be publicly available on Pubmed Central, in accordance with NIH guidelines for Sharing of Research Data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Commencing 24 months after the award initiation, all data will be deposited onto USC-provided OneDrive, with subsequent deposits occurring every six months thereafter.
Access Criteria: Public

REFERENCES:
- [Background] Pyatak EA, Carandang K, Rice Collins C, Carlson M. Optimizing Occupations, Habits, and Routines for Health and Well-Being With Lifestyle Redesign(R): A Synthesis and Scoping Review. Am J Occup Ther. 2022 Sep 1;76(5):7605205050. doi: 10.5014/ajot.2022.049269. PMID 36053733
- [Background] Pyatak EA, Carandang K, Vigen CLP, Blanchard J, Diaz J, Concha-Chavez A, Sequeira PA, Wood JR, Whittemore R, Spruijt-Metz D, Peters AL. Occupational Therapy Intervention Improves Glycemic Control and Quality of Life Among Young Adults With Diabetes: the Resilient, Empowered, Active Living with Diabetes (REAL Diabetes) Randomized Controlled Trial. Diabetes Care. 2018 Apr;41(4):696-704. doi: 10.2337/dc17-1634. Epub 2018 Jan 19. PMID 29351961